CLINICAL TRIAL: NCT00039299
Title: A Phase I Safety Study Of Xcellerate In Patients With Hormone Refractory Prostate Cancer
Brief Title: Biological Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: XCYTE-SPR-080011; UCLA-0111008; CDR0000069370 (Registry Identifier: PDQ (Physician Data Query)); XCYTE-XT002; NCI-G02-2075
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2003-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop tumor cells from growing. Treating a person's T cells in the laboratory and then reinfusing them may cause a stronger immune response and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of T-cell therapy in treating patients who have prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of activated autologous T cells (Xcellerate) therapy in patients with hormone-refractory prostate cancer.
* Determine the change in prostate-specific antigen (PSA) levels in patients treated with this therapy.
* Determine the effects on bone in patients treated with this therapy.

OUTLINE: This is a multicenter study.

Patients undergo leukapheresis to collect peripheral blood mononuclear cells (PBMC). PBMC are activated and expanded ex vivo by costimulation with antihuman CD3 and antihuman CD28 monoclonal antibodies covalently attached to superparamagnetic microbeads (Xcellerate). Xcellerate-activated T cells are reinfused on day 0.

Patients are followed weekly for 4 weeks and then monthly for 3 months.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Evidence of androgen-independent disease

    * Patient must have received prior primary hormonal therapy (e.g., orchiectomy or gonadotropin-releasing hormone analog with or without antiandrogen)
    * Demonstrated disease progression by any 1 of the following:

      * Elevated PSA level (at least 5 ng/mL) that has serially risen from baseline on 2 occasions at least 1 week apart
      * At least 1 new osseous lesion on bone scan
      * More than 25% increase in the sum of the products of the perpendicular diameters of all bidimensionally measurable sites of disease
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGPT no greater than 1.5 times ULN
* Hepatitis B surface antigen negative
* No active or chronic hepatitis B or C
* No other hepatic dysfunction that would preclude study

Renal:

* Creatinine less than 2.0 mg/dL
* Calcium less than 11 mg/dL
* No renal dysfunction that would preclude study
* No symptomatic hypercalcemia

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Pulmonary:

* No pulmonary disease requiring inhaled steroids or bronchodilators

Other:

* No history of HIV 1 or 2 or human T-cell lymphotrophic virus (HTLV) 1 or 2
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer
* No history of autoimmune disease (e.g., rheumatoid arthritis or multiple sclerosis)
* No other major organ system dysfunction
* No gastrointestinal, neurologic, or psychiatric dysfunction that would preclude study
* Human anti-mouse antibody negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent growth factors, interleukin, interferons, or cytokines

Chemotherapy:

* No prior chemotherapy or other systemic chemotherapy agent for prostate or any other cancer

Endocrine therapy:

* Prior aminoglutethimide allowed
* At least 4 weeks since prior flutamide
* At least 6 weeks since prior bicalutamide or nilutamide
* Concurrent luteinizing hormone-releasing hormone agonists should be continued
* No concurrent corticosteroids or dexamethasone
* No concurrent anti-androgens (e.g., flutamide, bicalutamide, or nilutamide)

Radiotherapy:

* At least 4 weeks since prior local radiotherapy
* No prior radiopharmaceutical therapy (e.g., strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium)
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* Prior ketoconazole or PC-SPES allowed
* At least 1 week since prior antibiotic, antifungal, or antiviral agents
* At least 4 weeks since other prior systemic therapy for prostate cancer (except bisphosphonates or hormonal therapy)
* At least 6 weeks since prior investigational drugs or devices
* No other concurrent therapy for this disease
* No concurrent participation in another clinical trial
* No concurrent bisphosphonates unless initiated prior to study
* No concurrent immunosuppressive drugs
* No other concurrent experimental therapies

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-03; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Pantuck, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States